CLINICAL TRIAL: NCT03773783
Title: Effectiveness of Treatment for Class II Malocclusions With the Button & Bead or Twin-block Functional Appliance: A Single Centre Randomised Clinical Trial
Brief Title: Study to Compare Two Functional Appliances for Class II Malocclusions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG_16-204
Record Dates: First submitted 2017-10-06; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Malocclusion, Angle Class II
Keywords: Myofunctional appliance
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin Block (Active Comparator): Twin Block appliance
  Interventions: Device: Twin Block appliance
- Button and Bead (Experimental): Button and Bead appliance
  Interventions: Device: Button and Bead appliance

INTERVENTIONS:
Device: Button and Bead appliance — Button and Bead appliance
  Arms: Button and Bead
Device: Twin Block appliance — Twin Block appliance
  Arms: Twin Block

SUMMARY:
A randomised controlled clinical trial to compare the effectiveness of two functional appliances in the correction of a Class II malocclusion. (Class II malocclusions are where upper front teeth bite significantly further forward in relation to lower front teeth).

Null hypothesis:

There is no significant difference between the Button & bead and Twin-block appliances with regard to time taken to reduce the overjet

DETAILED DESCRIPTION:
Background:

A functional appliance is a type of brace used to help correct a 'Class II' malocclusion. Class II malocclusions are where upper front teeth bite significantly further forward in relation to lower front teeth. A functional appliance is defined as a brace that engages upper and lower teeth and works mainly by posturing the lower jaw away from its normal position1. The functional appliance may either be removable or fixed in nature and of various designs.

Correction of a class II malocclusion can be commenced early i.e. before the age of 10 or during early adolescence when the patient is in a late mixed dentition / early permanent dentition. If correction is commenced early, this results in the need for a two phase treatment which involves functional appliance treatment in the first phase (age 7-10) followed by fixed appliances (+/- functional appliances) as an adolescent (age 11-16). If correction is started in early adolescence only one phase of treatment is required which involves a combination of functional and fixed appliances (age 11-16).

Early or delayed class II treatment has been studied by various researchers2-10. O'Brien et al7 concluded that there was no advantage of early treatment with Twin Block as compared to treatment started in adolescents. In fact, they reported significantly poorer occlusal outcomes as determined by the objective Peer Assessment Rating (PAR) index in those that had early treatment. In addition, they found that total duration of treatment, total attendances and total cost of treatment was significantly higher in the early treatment group. The average total duration of treatment for those that had early treatment was 968 days (phase 1 = 527 days and phase 2 = 435 days) compared to 744 days for those that had treatment as an adolescent only.

The most commonly used brace to correct class II malocclusions in the UK is a functional appliance (Twin Block design) 11.

The Button and Bead functional appliance has been developed and used successfully by Mr Spary (Consultant Orthodontist) for several years. However, there are no studies to date that have studied its effectiveness in correcting a class II problem. The Button and bead appliance appears to be quicker at reducing the overjet and preferred by patients as there is less mouth opening making the appliance more comfortable to wear. It is also two clear aligners, which are more aesthetic than the traditional twin block appliance. The button and bead appliance does not however allow arch expansion. This may necessitate another appliance prior to fixed appliance treatment or prolong fixed appliance treatment if expansion also needs to be carried out in that phase.

Objectives:

1. Primary objective:

   a. To compare the Button-&-bead and Twin-block appliances treatment duration for overjet reduction
2. Secondary objectives:

   1. To compare the Button-&-bead and Twin-block appliances dento-occlusal outcomes as measured by the Peer Assessment Rating (PAR)
   2. To compare patient compliance with the Button-&-bead and Twin-block appliances and identify causes for failure
   3. To compare the health economics of the Button-&-bead and Twin-block appliances (Cost of appliances, number of visits, number and cost of repairs and/or replacements)
   4. To compare the skeletal changes of the Button-&-bead and Twin-block appliances based on the Eastman analysis
   5. To compare changes in soft tissue profile as assessed by 3D photographs
   6. To assess changes in OHRQoL after overjet reduction with the Button-&-bead and Twin-block appliances
   7. To evaluate and compare patient satisfaction with the Button-&-bead and Twin-block appliances
3. Safety objective

   1. To evaluate the safety of the Button-&-Bead appliance relative to the Twin-Block appliance in terms of the occurrence of any device-related adverse- and side-effects (soft-tissue trauma, decalcification, dental caries, ingestion or aspiration of appliance).

ELIGIBILITY:
Inclusion Criteria:

* * Overjet ≥ 7mm

  * The normal overjet for a Caucasian population is in the range of 2-4mm. A functional appliance is used to allow for overjet reduction without extractions and/or to reduce the anchorage demands of the subsequent treatment with the Straight Wire Appliance (SWA). Clinically the overjet would need to be significantly increased for the treating clinician to consider the use of a functional appliance. Other similar studies have used an overjet of >6mm or ≥ 7mm. This study has elected for an initial overjet of ≥ 7mm to improve the studies external validity by making it more applicable to day-to-day clinical practice.
  * The initial overjet will be used to select patients. The majority of recent high level trials and systematic reviews that have provided a significant amount of the evidence base in the treatment of Class II malocclusions have defined subjects according to their initial overjet.

    * Age 10 to 14 years
  * This has been selected to match other studies relating to functional appliance treatment and reflect the most common clinical practice. The literature on functional appliance treatment has provided evidence that on average the enhancement of growth is small. Some studies on the timing of functional appliance treatment have suggested that pubertal growth is not a significant factor in the success of functional appliance treatment but it is well know and accepted that functional appliance treatment is assisted during periods of more rapid growth. Numerous studies have also found better co-operation and completion of treatment in younger patients (Banks 2004, KOB 2003a & 2003b)

    * Satisfactory Dental health
  * Patients must be dentally healthy and have a suitable level of oral health that would support orthodontic treatment, as per the British Orthodontic Society guidelines. They must have good oral hygiene with minimal gingivitis or periodontal disease, no dental caries or periapical pathology and no history of dento-alveolar trauma. This is judged by the investigator.

    * Willing to participate in study and provide informed consent

Exclusion Criteria:

* * No previous orthodontic treatment or premolar extractions

  * This is aimed at reducing any confounding factors within the study as these may affect the success of treatment.

    * No craniofacial syndrome (including Cleft patients)
  * This is aimed at reducing any confounding factors within the study as these conditions may affect the success of treatment. The treatment of this subgroup requires a multi-disciplinary team and is more complex. Their treatment pathway may vary from normal clinical practice.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in overjet reduction | Overjet measurement recorded at the start of treatment and at completion of functional appliance therapy 1 year later.
  How quickly the horizontal discrepancy between upper and lower incisor edges is reduced

SECONDARY OUTCOMES:
Change in Peer Assessment Rating (PAR) | PAR score will be Assessed from the start of treatment models and the end of fixed appliance study models ( 2 years later)
  PAR score change in terms of percentage and actual score
Drop out | No. of patients at the start of functional appliance therapy that do not wish to continue within the trial or do not finish functional appliance therapy within 18 months
  Percentage of patients dropping out of each arm of the trial
Skeletal changes | Cephalometric x-rays at start of treatment and at the end of treatment 1 year later
  Compare skeletal changes of landmarks in degrees and millimetres using cephalometric x-rays at various time points
3D soft tissue measures | 3D photographs at start of treatment and at the end of treatment (approx 1 year later)
  Measure changes in soft tissues using 3D photographs
Patient satisfaction | Patient satisfaction survey at study completion ( 1 year after treament started)
  Use of tailored patient satisfaction questionnaire to assess patient satisfaction with both appliances
Child related Oral health quality of life (OHRQoL) questionnaire | The patient ticked the applicable box for the 16 set questions from the standardised qualitative oral health questionairre. This was undertaken at the start of the trial and again at the end of functional appliance therapy ( approximately 1 year later)
  Changes in OHRQoL
Adverse events | Adverse events over the course of functional appliance treatment ( recorded at every visit and reviewed at 1 year)
  Adverse events: decalcification, dental caries, soft tissue trauma, ingestion or aspiration of appliance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham dental hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isaacson KG, Reed RT, Stephens CD. Functional orthodontic appliances. Oxford: Blackwell Scientific Publications; 1990.
- [Background] Tulloch JF, Phillips C, Proffit WR. Benefit of early Class II treatment: progress report of a two-phase randomized clinical trial. Am J Orthod Dentofacial Orthop. 1998 Jan;113(1):62-72, quiz 73-4. doi: 10.1016/S0889-5406(98)70277-X. PMID 9457020
- [Background] Keeling SD, Wheeler TT, King GJ, Garvan CW, Cohen DA, Cabassa S, McGorray SP, Taylor MG. Anteroposterior skeletal and dental changes after early Class II treatment with bionators and headgear. Am J Orthod Dentofacial Orthop. 1998 Jan;113(1):40-50. doi: 10.1016/S0889-5406(98)70275-6. PMID 9457018
- [Background] Ghafari J, Shofer FS, Jacobsson-Hunt U, Markowitz DL, Laster LL. Headgear versus function regulator in the early treatment of Class II, division 1 malocclusion: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 1998 Jan;113(1):51-61. doi: 10.1016/s0889-5406(98)70276-8. PMID 9457019
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of treatment for Class II malocclusion with the Herbst or twin-block appliances: a randomized, controlled trial. Am J Orthod Dentofacial Orthop. 2003 Aug;124(2):128-37. doi: 10.1016/s0889-5406(03)00345-7. PMID 12923506
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of early orthodontic treatment with the Twin-block appliance: a multicenter, randomized, controlled trial. Part 1: Dental and skeletal effects. Am J Orthod Dentofacial Orthop. 2003 Sep;124(3):234-43; quiz 339. doi: 10.1016/S0889540603003524. PMID 12970656
- [Background] O'Brien K, Wright J, Conboy F, Appelbe P, Davies L, Connolly I, Mitchell L, Littlewood S, Mandall N, Lewis D, Sandler J, Hammond M, Chadwick S, O'Neill J, McDade C, Oskouei M, Thiruvenkatachari B, Read M, Robinson S, Birnie D, Murray A, Shaw I, Harradine N, Worthington H. Early treatment for Class II Division 1 malocclusion with the Twin-block appliance: a multi-center, randomized, controlled trial. Am J Orthod Dentofacial Orthop. 2009 May;135(5):573-9. doi: 10.1016/j.ajodo.2007.10.042. PMID 19409339
- [Background] Nelson C, Harkness M, Herbison P. Mandibular changes during functional appliance treatment. Am J Orthod Dentofacial Orthop. 1993 Aug;104(2):153-61. doi: 10.1016/S0889-5406(05)81005-4. PMID 8338068
- [Background] Illing HM, Morris DO, Lee RT. A prospective evaluation of Bass, Bionator and Twin Block appliances. Part I--The hard tissues. Eur J Orthod. 1998 Oct;20(5):501-16. doi: 10.1093/ejo/20.5.501. PMID 9825553
- [Background] Thiruvenkatachari B, Sandler J, Murray A, Walsh T, O'Brien K. Comparison of Twin-block and Dynamax appliances for the treatment of Class II malocclusion in adolescents: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):144.e1-9; discussion 144-5. doi: 10.1016/j.ajodo.2010.01.025. PMID 20691354
- [Background] Chadwick SM, Banks P, Wright JL. The use of myofunctional appliances in the UK: a survey of British orthodontists. Dent Update. 1998 Sep;25(7):302-8. PMID 10478026